CLINICAL TRIAL: NCT06461819
Title: Safety of Dose Escalation in Definitive Hypofractionated Radiation Therapy With SPACEOAR TM for Patients With Low-to-intermediate Risk Localized Prostate Cancer (DESAR-L)
Acronym: DESAR-L
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Park, Won Park, M.D., Ph.D., Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2023-06-143
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Low-to-intermediate-risk Prostate Carcinoma

STUDY DESIGN:
Intervention Model Description: 2) Clinical study design
  -A single institution with a single group, a phase II study, Low- and medium-risk studies performed after biodegradable substance injection prostate cancer dose increase. We plan to evaluate grade 1 or higher rectal bleeding occurring within 3 years in patients who have received low -fractionation curative radiotherapy.
  3) Primary endpoint NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) V 5.0 Frequency of rectal bleeding of grade 1 or higher within 3 years
  4) Secondary endpoint
  1. Radiation therapy-related side effects other than rectal bleeding
  2. Side effects related to biodegradable material injection
  3. 5-year biochemical recurrence-free survival
  4. 5-year progression-free survival
  5. 5-year overall survival
  6. quality of life
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patient, candidate of definitive radiation treatment (Experimental): A single institution with a single group, a phase II study, Low- and medium-risk studies performed after biodegradable substance injection prostate cancer dose increase.
  Interventions: Radiation: Low- and medium-risk studies performed after biodegradable substance injection prostate cancer dose increase.

INTERVENTIONS:
Radiation: Low- and medium-risk studies performed after biodegradable substance injection prostate cancer dose increase. — this researcher used a biodegradable material injection technique. after subdivision radical received radiation therapy We plan to conduct a phase II clinical study to evaluate the safety of prostate cancer patients.

SUMMARY:
A single institution with a single group, a phase II study, low- and medium-risk studies performed after biodegradable substance injection prostate cancer dosage increase. The investigator plans to evaluate grade 1 or higher rectal bleeding occurring within 3 years in patients who have received low -fractionation curative radiotherapy.

DETAILED DESCRIPTION:
In prostate cancer, radiation therapy for curative purposes can be used regardless of stage if there is no distant metastasis. For prostate cancer patients with low-and medium risk, radiotherapy is recommended as standard treatment along with surgery. In randomized prospective studies to investigate the therapeutic effect of dose escalation over 70 Gy during radiation therapy, increasing dose showed a significant reduction in biochemical failure. When the dose is increased, the risk of side effects (digestive system, urinary system) in surrounding normal tissues increases, and intensity modulated radiation therapy (IMRT) or image-guided radiation therapy (IGRT) Application could reduce the probability of side effects. Prostate cancer is a carcinoma characterized by slow growth, and the estimated α/β ratio is 1.5, which is smaller than surrounding normal tissues such as the bladder (4.0) and the rectum (3.9). Therefore, efforts to obtain therapeutic gain through hypofractionated radiation therapy have been attempted using three-dimensional conformal radiotherapy (3D-CRT) and IMRT. In particular, in the CHHIP trial11 announced in 2016, normal division Radiation therapy (74 Gy, 37 splits ) and As a result of comparing low-fractionation radiation therapy (60 Gy, 20 fractions ), there was no significant difference in the 5-year biochemical or clinical recurrence -free survival rate of low-fractionation radiation therapy, it was also reported that there was no difference in rectal and bladder side effects. However, rectal and bladder side effects of grade 2 or higher were 11.9% and 11.7 % during one-time 3 Gy low-fractionated radiotherapy, respectively. The low-fractionated radiotherapy dose is 81 Gy, which is the recommended normal fractionated radiotherapy dose when using IMRT. It can be said that there is a high possibility of showing inferior treatment results in long-term follow-up results because the biological effective dose is lower than that of 'ideal'. (Table 1)

* Table 1 . Biological Equivalent Dose by Radiation Therapy Policy(2-Gy fraction) comparison
* Protocol: EQD2 (Gy) (α/β=1.5)
* Low-fraction radiation therapy(70 Gy, 28 sessions): 80.0 Gy
* Conventional fractionation radiation therapy(74 Gy, 37 times): 74 Gy
* CHHIP trial(60 G y, 20 times): 77. 14 Gy
* study design dose(64 Gy, 20 times): 85.94 Gy *EQD2, equivalent dose in 2-Gy fractions

Recently, a method was devised to increase the distance between prostate and rectum by injecting hydrogel between prostate and rectum to minimize rectal dose even when performing high-dose radiotherapy to prostate. In particular, a biodegradable material ( SpaceOAR (hydrogel)) that is absorbed into the body after a certain period of time has been developed, and radical radiation therapy is performed. It is currently being used in prostate cancer patients. It is judged possible to try to increase the radiation dose because the side effects can be reduced by reducing the rectal dose during radical radiation treatment through biodegradable material injection. So far, studies evaluating the side effects of treatment according to increased radiation dose after injection of biodegradable materials are very limited.

Therefore, the investigator uses a biodegradable material injection technique follows by subdivision radical received radiation therapy. The investigator plans to conduct a phase II clinical study to evaluate the safety of prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer patients confirmed histopathologically within 6 months prior to study enrollment
2. Low-risk and medium- risk groups in terms of risk Prostate cancer patients (primary stage T2c or less, Grade group 3 or less, If PSA is less than 20ng/ml)
3. Adults over 20 years of age
4. Whole body performance ECOG 0-1
5. SpaceOAR Patients who consented to the procedure and the clinical study

Exclusion Criteria:

1. Prostatectomy, Patients with a history of lower pelvic surgery including rectal cancer surgery
2. primary cancer Patients with posterior extracapsular extension
3. Medically biodegradable substances such as bleeding predisposition Patients for whom infusion is not appropriate
4. Biodegradable material Patients who failed infusion
5. Patients with a history of previous pelvic radiation therapy
6. Patients with distant metastasis and intrapelvic lymph node metastasis
7. Patients who have undergone or are scheduled to undergo hormone therapy

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer patients confirmed histopathologically within 6 months prior to study enrollment
Enrollment: 33 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) V 5.0 Frequency of rectal bleeding of grade 1 or higher within 3 years | 5 years after radiation therapy of each participant
  NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) V 5.0

SECONDARY OUTCOMES:
Radiation therapy-related side effects other than rectal bleeding | 5 years after each participant's end of radiation therapy after SpaceOAR hydrogel injection
  Radiation therapy-related side effects other than rectal bleeding
Side effects related to biodegradable material injection | 5 years after radiation therapy of each participant
  Side effects related to biodegradable material injection
5-year biochemical recurrence-free survival | 5 years after radiation therapy of each participant
  5-year biochemical recurrence-free survival
5-year progression-free survival | 5 years after radiation therapy of each participant
  5-year progression-free survival
5-year overall survival | 5 years after radiation therapy of each participant
  5-year overall survival
quality of life in every aspect of life | 5 years after radiation therapy of each participant
  quality of life using Questionnare EPIC ( Extended Prostate Cancer Index Composite)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- See also: SpaceOAR™ Hydrogel is Associated with Lower Rectal Toxicity and Higher Bowel Quality of Life in Late Follow-up: Systematic Review & Meta-Analysis — https://www.bostonscientific.com/content/dam/bostonscientific/spaceoar/vue/infographic-spaceoar-hydrogel-meta-analysis.pdf